CLINICAL TRIAL: NCT03068715
Title: Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression (SAINT-TRD)
Acronym: aTBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistaant Professor, Psychiatry & Behavioral Sciences, Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Blinded-33797
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Treatment Resistant Depression
Keywords: transcranial magnetic stimulation; theta burst
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TBS-DLPFC (Experimental): The active group will receive theta-burst TMS stimulation.
  Interventions: Device: Active TBS-DLPFC; Device: Open label TBS-DLPFC
- Sham TBS-DLPFC (Sham Comparator): The sham group will receive sham theta-burst TMS stimulation.
  Interventions: Device: Sham TBS-DLPFC; Device: Open label TBS-DLPFC

INTERVENTIONS:
Device: Active TBS-DLPFC — Participants in the active stimulation group will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator.
  Arms: Active TBS-DLPFC
Device: Sham TBS-DLPFC — The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham TBS-DLPFC
Device: Open label TBS-DLPFC — All patients will have the option to receive active, open label aTBS treatment after the 1-month mark, following the blinded phase.
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator or Nexstim TMS device.

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for treatment-resistant depression. In a double-blind fashion, half the participants will receive accelerated theta-burst stimulation while half will receive sham treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been effective in real world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session, 5 days per week, for 4-8 weeks). Recently, researchers have pursued modifying the treatment parameters to reduce treatment times with some preliminary successes. This study aims to further modify the parameters to create a more rapid form of the treatment and look at the change in neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 22 to 80 years of age.
* Able to provide informed consent.
* Diagnosed with Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE).
* Participants may currently be on a stable and adequate dose of SSRI antidepressant therapy. Participants may choose to not be on antidepressant therapy for the study duration, or to be switched from other classes to a medication from the SSRI class.
* Participants may also have a history of intolerance to at least 2 antidepressant medications. These patients with the intolerance history will not be required to be currently taking an antidepressant medication.
* Participants must qualify as "Moderately Treatment Refractory" or "High Treatment Refractory" using the Maudsley staging method.
* Meet the threshold on the total HAMD17 score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total MADRS score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total BDI-II score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* In good general health, as ascertained by medical history.
* If female, a status of non-childbearing potential or use of an acceptable form of birth control. The form of birth control will be documented at screening and baseline.
* Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
* Female that is pregnant or breastfeeding.
* Female with a positive pregnancy test at participation.
* Total HAMD17 score of < 20 at the screen or baseline visits.
* Total MADRS score of < 20 at the screen or baseline visits.
* Total BDI-II score of < 20 at the screen or baseline visits.
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine dependence, at screening or within six months prior to screening.
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening.
* Considered at significant risk for suicide during the course of the study.
* Cognitive impairment (as noted by previous diagnoses-including dementia).
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
* Current (or chronic) use of opiates.
* History of epilepsy.
* History of rTMS exposure.
* History of any implanted device or psychosurgery for depression.
* Any history of ECT (greater than 8 sessions) without meeting responder criteria
* History of shrapnel or metal in the head or skull.
* "Low Treatment Refractory" using the Maudsley staging method.
* History of cardiovascular disease or cardiac event.
* History of OCD.
* History of autism spectrum disorder.
* History of intractable migraine
* History of independent sleep disorder.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2021-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396
- [Derived] Batail JM, Xiao X, Azeez A, Tischler C, Kratter IH, Bishop JH, Saggar M, Williams NR. Network effects of Stanford Neuromodulation Therapy (SNT) in treatment-resistant major depressive disorder: a randomized, controlled trial. Transl Psychiatry. 2023 Jul 3;13(1):240. doi: 10.1038/s41398-023-02537-9. PMID 37400432
- [Derived] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TBS-DLPFC: The active group will receive theta-burst TMS stimulation.
  Active TBS-DLPFC: Participants in the active stimulation group will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator.
  Open label TBS-DLPFC: All patients will have the option to receive active, open label aTBS treatment after the 1-month mark, following the blinded phase.
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator or Nexstim TMS device.
- Sham TBS-DLPFC: The sham group will receive sham theta-burst TMS stimulation.
  Sham TBS-DLPFC: The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Open label TBS-DLPFC: All patients will have the option to receive active, open label aTBS treatment after the 1-month mark, following the blinded phase.
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator or Nexstim TMS device.
Period: Overall Study
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — No longer met inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active TBS-DLPFC: The active group will receive theta-burst TMS stimulation.
  Active TBS-DLPFC: Participants in the active stimulation group will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator.
- Total: Total of all reporting groups
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 49 [27 to 73] | 52 [30 to 72] | 51 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 13 | 25
  Asian | 2 | 1 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Years of education [Mean (Full Range); unit: years] | 17 [13 to 27] | 17 [12 to 30] | 17 [12 to 30]
Currently employed [Count of Participants; unit: Participants] | 7 | 6 | 13
Duration of illness [Mean (Full Range); unit: years] | 30 [1 to 62] | 23 [1 to 56] | 26 [1 to 62]
Duration of current depressive episode [Mean (Full Range); unit: years] | 8 [0 to 53] | 10 [1 to 46] | 9 [0 to 53]
ATHF adequate antidepressant trials, lifetime [Mean (Full Range); unit: number of lifetime antidepressant trials] | 5 [3 to 9] | 5 [0 to 8] | 5 [0 to 9]
ATHF adequate augmentation trials, lifetime [Mean (Full Range); unit: number of lifetime augmentation trials] | 1 [0 to 4] | 1 [0 to 3] | 1 [0 to 4]
ATHF adequate antidepressant trials, current episode [Mean (Full Range); unit: number of current antidepressant trials] | 2 [0 to 4] | 1 [0 to 3] | 2 [0 to 4]
ATHF adequate augmentation trials, current episode [Mean (Full Range); unit: number of current augmentation trials] | 1 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
Maudsley Staging Method Score [Mean (Full Range); unit: score on a scale] — The Maudsley Staging Method (MSM) is a points-based staging model incorporating 3 factors: treatment, severity of illness, and duration of presenting episode. The overall level of resistance estimated using this model varies from minimal resistance (score of 3) to severe resistance (score of 15).
  score on a scale | 9 [6 to 12] | 9 [5 to 13] | 9 [5 to 13]
Baseline MADRS overall score [Mean (Full Range); unit: score on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS), is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Overall scores above 34 indicate severe depression.
  score on a scale | 31 [25 to 38] | 35 [24 to 50] | 33 [24 to 50]
Baseline HAM-6 score [Mean (Full Range); unit: score on a scale] — The Hamilton Depression Rating Scale (HDRS, also known as Ham-D) is the most widely used clinician-administered depression assessment scale.
  Scores can range from 0 to 22. Higher scores represent higher depression severity.
  score on a scale | 14 [11 to 17] | 15 [11 to 18] | 15 [11 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Score From Pre-treatment to 1-month Post-treatment.
Description: A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.
Time Frame: Pretreatment (baseline), 1-month post-treatment
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change in MADRS score
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 14 | 15
percent change in MADRS score | -53 (35) | -11 (29)
Statistical Analysis 1: Comparison: Active TBS-DLPFC vs Sham TBS-DLPFC; MADRS scores were assessed with generalized linear mixed models (GLMM) that used Satterthwaite approximation of degrees of freedom and robust estimation of coefficients to handle violations of model assumptions. Fixed effects of time, treatment group (sham vs. active) and their interaction were assessed; Test type: Superiority — We assessed the superiority of active over sham; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Percentage Change in the Hamilton Rating Scale for Depression (HAMD-17)
Description: A provider administered questionnaire used to assess remission and recovery from depression. The HAMD-17 is a 17-item questionnaire to assess depression severity. Each item is scored from 0-4, with higher scores representing increasing depression severity.
Time Frame: pre-treatment (baseline) to 1-month post-treatment
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change in HAM-17 score
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 14 | 15
percent change in HAM-17 score | -52 (29) | -12 (27)
Statistical Analysis 1: Comparison: Active TBS-DLPFC vs Sham TBS-DLPFC; HDRS-17 scores were assessed with generalized linear mixed models (GLMM) that used Satterthwaite approximation of degrees of freedom and robust estimation of coefficients to handle violations of model assumptions. Fixed effects of time, treatment group (sham vs. active) and their interaction were assessed; Test type: Superiority — We assessed the superiority of active over sham; p = 0.001, Mixed Models Analysis

3. Secondary Outcome: Change in the Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide assessment developed by multiple institutions including Columbia University. Participants were asked a series of 6 yes or no questions. Yes answers indicate more suicidal ideation. Here we report a count of participants with an increase, decrease or no change in suicidal ideation.
Time Frame: Pretreatment (baseline) to immediately post-treatment (day 8).
Population: Participants with available data are included in this analysis. Only participants with paired data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 8 | 6
Participants
  Increased | 0 | 0
  Decreased | 6 | 1
  No Change | 2 | 5

4. Secondary Outcome: Change in the Hamilton Rating Scale for Depression (HAM-6) Score
Description: The Hamilton Depression Rating Scale (HDRS, also known as Ham-D) is the most widely used clinician-administered depression assessment scale.
  The Ham-6 version consists of 6 items assessing for: mood, guilt, general somatic symptoms, work and activities, anxiety and slowness of thought and speech). Each item is scored on a scale of 0 to 4, except for the somatic symptoms item, which is scored 0 to 2. On the HAM-6 there can be a total score of 22. Higher scores represent higher depression severity. Here, we report a count of participants with an overall increase, decrease or no change in total HAM-6 score.
  Participants with an increase in total score (row 3) would signify a worse outcome than participants with a decrease in total score.
Time Frame: Baseline (pre-treatment) and at 1-month post-treatment
Population: Participants with available data are included in this analysis. Only participants with paired data are included.
  Scores are marked as a change from baseline if the difference is greater than 1 point.
Measure: Count of Participants; unit: Participants
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 11 | 10
Participants
  Decreased | 8 | 3
  No Change | 2 | 6
  Increased | 1 | 1

5. Secondary Outcome: Percentage Change in the Hamilton Rating Scale for Depression (HAMD-17)
Description: The Hamilton Depression Rating Scale (HDRS, also known as Ham-D) is the most widely used clinician-administered depression assessment scale.
  The Ham-17 version consists of 17 items assessing for: mood, guilt, general somatic symptoms, work and activities, anxiety and slowness of thought and speech. Each item is scored on a scale of 0 to 4, except for the somatic, sleep and insight items which are scored 0 to 2. On the HAM-17 there can be a total score of 22. Higher scores represent higher depression severity.
Time Frame: Pre-treatment (baseline) to immediately post-treatment (day 8).
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 14 | 15
percent change in score | -59 (31) | -20 (22)
Statistical Analysis 1: Comparison: Active TBS-DLPFC vs Sham TBS-DLPFC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — We assessed the superiority of active over sham; p = 0.001, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline Functional Connectivity to Immediate Post-treatment
Description: We quantified the functional connectivity change between the subcallosal cingulate to the default mode network and within the default mode network using baseline and immediate post-treatment MRI scans. We report below, changes of functional connectivity (Fisher's Z score of Pearson correlation coefficient for each pair of ROIs) from immediately post-treatment (day 8) to baseline.
Time Frame: Pretreatment (baseline) to immediately post-treatment (day 8).
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 13 | 12
Z-score
  lsgACC_lDMN | 0.071 (0.242) | 0.025 (0.301)
  lDMN_rDMN | -0.069 (0.330) | 0.117 (0.565)
Statistical Analysis 1: Comparison: Active TBS-DLPFC; Functional connectivity between lsgACC_lDMN in participants receiving active iTBS; Test type: Superiority — FC was calculated as the correlation (Pearson) of the activity pattern across time between ROIs. All Pearson correlation coefficients were then transformed into Fisher's Z score for further analysis. sgACC (BA25) was defined by Brodmann areas (BA). The 4 nodes of DMN were extracted from the Multi-Subject Dictionary Learning (MSDL) atlas; p = 0.308, t-test, 2 sided; Paired-t test was used for the statistics
Statistical Analysis 2: Comparison: Sham TBS-DLPFC; Functional connectivity between lsgACC_lDMN in participants receiving sham iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.778, t-test, 2 sided; Paired t-test was used for the statistics
Statistical Analysis 3: Comparison: Active TBS-DLPFC; Functional connectivity between lDMN_rDMN in participants receiving active iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.468, t-test, 2 sided; Paired t-test was used for the statistics
Statistical Analysis 4: Comparison: Sham TBS-DLPFC; Functional connectivity between lDMN_rDMN in participants receiving sham iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.486, t-test, 2 sided; Paired t-test was used for the statistics

7. Secondary Outcome: Change From Baseline Functional Connectivity to 1-month Post-treatment
Description: We will assess functional connectivity as seen on resting state fMRI, between the subcallosal cingulate to the default mode network and within the default mode network. We report below, changes of functional connectivity (Fisher's Z score of Pearson correlation coefficient for each pair of ROIs) from post-treatment(1m) to baseline.
Time Frame: Pretreatment (baseline) to 1-month post-treatment
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 13 | 11
Z-score
  lsgACC_lDMN | 0.090 (0.287) | -0.163 (0.258)
  lDMN_rDMN | -0.039 (0.702) | -0.056 (0.388)
Statistical Analysis 1: Comparison: Active TBS-DLPFC; Functional connectivity between lsgACC_lDMN in participants receiving active iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.447, t-test, 2 sided; Paired t-test was used for the statistics
Statistical Analysis 2: Comparison: Sham TBS-DLPFC; Functional connectivity between lsgACC_lDMN in participants receiving sham iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.115, t-test, 2 sided; Paired t-test was used for the statistics
Statistical Analysis 3: Comparison: Active TBS-DLPFC; Functional connectivity between lDMN_rDMN in participants receiving active iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.546, t-test, 2 sided; Paired t-test was used for the statistics
Statistical Analysis 4: Comparison: Sham TBS-DLPFC; Functional connectivity between lDMN_rDMN in participants receiving sham iTBS; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.607, t-test, 2 sided

8. Secondary Outcome: Change in Baseline Heart Rate Variability to 1-month Post-treatment
Description: Heart rate variability measures will be compared pre-treatment and 1-month post-treatment.
Time Frame: Pretreatment to 1-month post-treatment
Population: Smaller than the total number of participants because some did not have data collected for this measure at either timepoint.
Measure: Mean (Standard Error); unit: SDNN in milliseconds
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 10 | 9
SDNN in milliseconds | 46.609 (25.262) | -26.670 (36.464)
Statistical Analysis 1: Comparison: Active TBS-DLPFC vs Sham TBS-DLPFC; We conducted a linear mixed models analysis, with a focus on the interaction term. No power analysis for this measure because number of participants was determined by other primary study aims; Test type: Superiority; p < 0.05, Mixed Models Analysis — Not adjusted for multiple comparisons at this time; We were interested in the interaction between treatment condition and timepoint; P value of the interaction = 0.110

9. Secondary Outcome: Change in Baseline Heart Rate Variability to Immediate Post-treatment
Description: Heart rate variability measures will be compared pre-treatment and immediately post-treatment.
Time Frame: Pretreatment to immediate post-treatment (day 8).
Population: Data from 18 participants analyzed. Smaller than the total number of participants for this study because some participants were missing one or both of the timepoints needed for this variable.
Measure: Mean (Standard Error); unit: SDNN in milliseconds
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
Number analyzed (Participants) | 9 | 9
SDNN in milliseconds | 16.226 (15.245) | -31.159 (35.258)
Statistical Analysis 1: Comparison: Active TBS-DLPFC vs Sham TBS-DLPFC; We used a linear mixed models analysis, with the fixed factors being treatment group and timepoint; Test type: Superiority — The SDNN (the standard deviation of the RR intervals) was recorded using ECG. It was not necessary to conduct a power analysis for this measure because the number of participants in the study was based on other considerations (primary treatment goals of the study); p < 0.05, Mixed Models Analysis — For reporting purposes here the p value was not adjusted for multiple comparisons; We were interested in the significance of the interaction between treatment group and timepoint; P value of the interaction = 0.245

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Active TBS-DLPFC | Sham TBS-DLPFC
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 12/14 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active TBS-DLPFC (N=14) | Sham TBS-DLPFC (N=15)
Fatigue (General disorders) | 8 | 8
Neck/back discomfort (Musculoskeletal and connective tissue disorders) | 7 | 5
Discomfort at treatment site (General disorders) | 5 | 2
Post-SAINT headache (Nervous system disorders) | 8 | 2
Anxiety (Nervous system disorders) | 4 | 3
Dental issues (General disorders) | 1 | 0
Jaw discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Polydipsia (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Data analysis for secondary outcome measures 3 (Change in C-SSRS score) and 4 (Change in HAM-6 score) are considered to be under powered, due to small number of subjects having available data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03068715/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT03068715/SAP_000.pdf